CLINICAL TRIAL: NCT07312292
Title: Radioembolization With Intra-arterial Angiotensin II to Improve Tumor-absorbed Dose
Brief Title: Radioembolization With Intra-arterial Angiotensin II to Improve Tumor-absorbed Dose (RADIANT)
Acronym: RADIANT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Niek Wijnen (Other)
Collaborators: PAION Deutschland GmbH (Industry)
Responsible Party: Sponsor-Investigator, Niek Wijnen, MD, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24U-0008; 2025-521870-33-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-16; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Liver Cancer (Locally Advanced or Metastatic); Liver Cancer Adult
Keywords: Radioembolization; Angiotensin II; yttrium-90
MeSH Terms: conditions — Liver Neoplasms; Neoplasm Metastasis; Carcinoma, Hepatocellular | interventions — Angiotensin II; Giapreza

STUDY DESIGN:
Intervention Model Description: The RADIANT study is a single-center, single-arm, phase II interventional clinical trial designed to evaluate the effect of intra-arterial angiotensin II (AT-II) infusion on tumor selectivity during yttrium-90 (⁹⁰Y) radioembolization in patients with primary or metastatic liver tumors.
  Each participant serves as their own control by comparing tumor-to-non-tumor ratio (TNR) measurements obtained during the standard radioembolization work-up (without AT-II) to measurements obtained during the therapeutic radioembolization procedure (with AT-II infusion).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radioembolization with intra-arterial angiotensin II (Experimental): Single-arm study in which all participants undergo standard yttrium-90 (⁹⁰Y) radioembolization for primary or metastatic liver tumors. During the therapeutic radioembolization procedure, angiotensin II is administered intra-arterially immediately prior to ⁹⁰Y glass microsphere injection at each arterial injection position.
  Interventions: Drug: Angiotensin II (Giapreza®); Radiation: Yttrium-90 radioembolization

INTERVENTIONS:
Drug: Angiotensin II (Giapreza®) — Angiotensin II is administered intra-arterially into the hepatic artery during the therapeutic radioembolization procedure. After confirmation of correct microcatheter position, angiotensin II is infused at a dose of 10 µg/min for 100 seconds, immediately followed by injection of yttrium-90 glass microspheres (TheraSphere®).
  In participants with multiple arterial injection positions, angiotensin II is administered at each injection position. In cases where whole-liver treatment is performed in two separate sessions, angiotensin II is administered during both treatment sessions.
  Dose: 10 µg/min Duration of Administration: 100 seconds per injection position Route of Administration: Intra-arterial (hepatic artery)
Radiation: Yttrium-90 radioembolization — Selective intra-arterial administration of yttrium-90 glass microspheres for the treatment of primary or metastatic liver tumors, performed according to standard clinical protocol.

SUMMARY:
This clinical trial will test whether a short infusion of a drug called angiotensin II can make a liver cancer treatment work better. The drug is given directly into the artery that supplies blood to the liver, right before a treatment called yttrium-90 (90Y) radioembolization.

The main questions it aims to answer are:

* Does angiotensin II help more of the radioactive beads reach the tumor and less reach the healthy parts of the liver?
* Is it safe to add angiotensin II to the standard radioembolization treatment? What will participants do?
* First visit (work-up): Participants will have the standard preparation for radioembolization. A small test dose of radioactive tracer (99mTc-MAA) will be injected into the liver through an artery. On the same day, a SPECT/CT scan will be performed to see how the tracer distributes in the liver and if there are depositions outside the liver. If everything looks good, the participant will return for treatment in 2-3 weeks.
* Second visit (treatment): Participants will receive the actual radioembolization treatment. At each injection site in the liver, first angiotensin II is administered, immediately followed by the injection of the radioactive beads (90Y microspheres). If the treatment requires injections in multiple locations, the participant will receive angiotensin II at each spot.
* After treatment: Participants will receive a PET/CT scan so the research team can see where the radioactive beads went. This will be compared to the distribution of the radioactive tracer (99mTc-MAA) from the first SPECT/CT scan (performed without angiotensin II) to measure how much angiotensin II helped target the tumor.

All monitoring (including blood pressure, heart rate, oxygen saturation, and breathing rate) takes place during the procedure as part of routine care, and there are no extra hospital visits beyond what is normally required for radioembolization.

ELIGIBILITY:
Inclusion criteria:

* Patients diagnosed with primary or metastatic liver tumors (any histological type).
* A clinical indication for radioembolization.
* Liver tumors with a diameter ≥ 2 cm.
* Age ≥ 18 years.
* Competent and able to provide own informed consent (no legally designated representative).
* Written informed consent.

Exclusion criteria:

* Any serious comorbidity preventing the safe administration of AT-II. This includes:

  1. Uncontrolled hypertension.
  2. Treatment with ≥ 3 antihypertensive drugs.
  3. Arterial (cerebro-)vascular or venous thromboembolic event within the past 6 months.
* Current use of angiotensin-converting enzyme (ACE) inhibitors.
* Current use of angiotensin II receptor blockers (ARBs).
* Known hypercoagulable state (i.e., thrombophilia).
* History of severe peripheral vascular disease.
* Known hypersensitivity to the active substance in Giapreza: angiotensin II.
* Known hypersensitivity to any of the excipients in Giapreza: mannitol, sodium hydroxide or hydrochloric acid.
* Any serious and/or chronic liver disease preventing the safe administration of radioembolization.
* Uncorrectable extrahepatic deposition of scout dose activity; activity in the falciform ligament, portal lymph nodes, and gallbladder is accepted.
* Pregnancy or breastfeeding.
* Body weight over 150 kg (because of maximum table load).
* Known severe allergy to intravenous contrast fluids.
* Participation in another investigational study which may compromise any endpoint of the study.
* Any other significant comorbidity or medical condition that may compromise the safety of radioembolization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Tumor-to-non-tumor ratio (TNR) improvement factor | From work-up procedure (baseline ⁹⁹ᵐTc-MAA SPECT/CT) to post-treatment imaging following radioembolization (⁹⁰Y PET/CT), within approximately 2-3 weeks.
  The tumor-to-non-tumor ratio (TNR) improvement factor is defined as the ratio of the TNR measured after yttrium-90 (⁹⁰Y) radioembolization with intra-arterial angiotensin II infusion to the TNR measured during the standard work-up procedure without angiotensin II.
  TNR after treatment is quantified using post-radioembolization ⁽⁹⁰Y⁾ PET/CT imaging. Baseline TNR is quantified using technetium-99m macroaggregated albumin (⁹⁹ᵐTc-MAA) SPECT/CT imaging obtained during the work-up procedure. TNR values represent the ratio of microsphere activity concentration in tumor tissue relative to non-tumorous liver parenchyma.

SECONDARY OUTCOMES:
Safety and toxicity of intra-arterial angiotensin II infusion combined with radioembolization | From start of angiotensin II infusion during the therapeutic procedure until completion of post-procedural monitoring (up to 1 hour after the procedure).
  Assessment of adverse events related to intra-arterial angiotensin II infusion in combination with yttrium-90 radioembolization. Adverse events are graded according to the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.
  Safety evaluation includes hemodynamic effects (e.g., changes in blood pressure, heart rate), procedural complications, and any other treatment-emergent adverse events.
Technical success of intra-arterial angiotensin II administration | During the therapeutic radioembolization procedure.
  Technical success is defined as the successful intra-arterial administration of angiotensin II at a dose of 10 µg/min for 100 seconds at the intended hepatic arterial injection position(s), followed immediately by delivery of yttrium-90 glass microspheres.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Utrecht, Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Patient privacy

REFERENCES:
- [Result] van den Hoven AF, Smits ML, Rosenbaum CE, Verkooijen HM, van den Bosch MA, Lam MG. The effect of intra-arterial angiotensin II on the hepatic tumor to non-tumor blood flow ratio for radioembolization: a systematic review. PLoS One. 2014 Jan 17;9(1):e86394. doi: 10.1371/journal.pone.0086394. eCollection 2014. PMID 24466071